CLINICAL TRIAL: NCT04134572
Title: Registry of Ollier Disease and Maffucci Syndrome That Collects Clinical, Functional, Genetic, Genealogical, Imaging, Surgical, Treatment, Quality of Life Data. Data is Linked to Patients' Biological Samples, When Available
Brief Title: Registry of Ollier Disease and Maffucci Syndrome
Acronym: ROM
Status: Recruiting | Type: Observational
Sponsor: Luca Sangiorgi (Other)
Responsible Party: Sponsor-Investigator, Luca Sangiorgi, Head of Departement of Rare Skeletal Disorders, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: 378/2017
Record Dates: First submitted 2019-10-14; First posted 2019-10-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Ollier Disease; Maffucci Syndrome
Keywords: Disease Registry; Natural History Study; Disease Evolution
MeSH Terms: conditions — Enchondromatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Biospecimen Retention: Samples With DNA — Whole peripheral blood, DNA, lymphocytes, tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ollier Disease and Maffucci Syndrome patients: The group comprises all patients affected by Ollier Disease and Maffucci Syndrome.

SUMMARY:
REM is a retrospective and prospective registry, finalized to care and research. It is articulated in main sections - strongly related and mutually dependent on each other - corresponding to different data domains: personal information, clinical data, genetic data, genealogical data, surgeries, etc..

This approach has been individuated in order to corroborate and integrate data from different resources and aspects of the diseases and to correlate genetic background and phenotypic outcomes, in order to better investigate diseases pathophysiology. Due to legal requirements, institutional directives and organizational issues, we are unable to include individuals residing outside Italy in the registry at this time. We are currently engaged in the preparation of a recruitment process for individuals residing outside Italy.

DETAILED DESCRIPTION:
The traditional method of collecting patient information is often chaotic, inconvenient and sometimes even unsafe, particularly when dealing with rare diseases. In 2017, the need to simplify the diagnostic process and to overcome the difficulties of data storage and analysis, led to the suggestion of implementing the Registry of Ollier Disease and Maffucci Syndrome (ROM).

The ROM relies on an IT platform named Genotype-phenotype Data Integration platform - GeDI. This solution, realized by a collaboration among Medical Genetic Department and a local software-house (Dilaxia Spa), is a General Data Protection Regulation (GDPR)-compliant, multi-client, web-accessible system and it has been designed according to current medical informatics standards (Orphanet code, ICD-10, Human Genome Variants Society, Findability Accessibility Interoperability Reusability Principles). GeDI is continuously implemented to improve management of persons with Ollier Disease and Maffucci Syndrome and to help researchers in analyzing collected information. ROM is articulated in main sections:

* Personal data: it comprises general information, birth details and residence data;
* Patient data: including the patients internal code, the hospital code and other patient details;
* Diagnostic Process: the diagnosis, the status (affected, suspected, etc.), age at diagnosis, comorbidities, allergies, etc.;
* Genogram: a tool for designing the family transmission of the disease, alongside information on the disease status of all relatives included;
* Clinical events: it records a long list of signs and symptoms of Ollier Disease and Maffucci Syndrome as well as several additional items to describe the disease
* Genetic Analysis and Alteration: including analytical technique, sample information, analysis duration, etc. This section also comprises detailed information on any detected pathological variants (e.g. gene, international reference, DNA change, protein change, genomic position, etc.);
* Visits: this section includes visit type (genetic, orthopedic, rehabilitation, pediatric, etc.), the date of the visit, prescriptions, imaging, etc.;
* Treatments: this section comprises information of a wide range of treatments including pharmacological, devices, supplements, and other treatments such as psychological, nutritional, etc.;
* Surgeries: this section contains information on the type of surgeries, the age of the patients, the site/localization of the procedures, etc.
* Documents: this repository allow us to store all types of documents (radiological reports, imaging, consents, clinical reports, etc.);
* Consents: this section provides a comprehensive overview of all consents collected, including the collection date;
* Samples: this section includes information on the samples, like the type, date of collection, etc.
* PROs: this section collects information on patients reported outcomes such as the quality of life or ABC scale.

ELIGIBILITY:
Inclusion Criteria:

* All patients affected by Ollier Disease and Maffucci Syndrome

Exclusion Criteria:

* Any condition unrelated to Ollier Disease and/or Maffucci Syndrome

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients affected by Ollier Disease and Maffucci Syndrome
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-01-16 (Actual); Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Natural History and Epidemiology in terms of clinical, genetic and functional evaluation | 25 years
  To maintain an established registry in order to assess epidemiology and natural history.
  Collection of:
  1. physical examinations data: assessment of severity of the disease
  2. orthopedic and functional data: stature (cm), weight (kg), number and localization of sites affected by enchondromas, site of malignant transformation, definition of deformities (localization and number), definition of limitations (localization and number)
  3. surgical procedures: type, number and site of surgeries disease-related and age at surgeries
  4. genetics background: target gene, type of mutation, type of variant detected, clinical significance
  5. family history: inheritance in maternal or paternal line
  6. treatment information: pharmacological, devices, supplements, and other treatments
  Clinical, orthopedic, surgical, treatment and functional features are updated at each follow up. Clinical reports, medical charts and imaging are the primary sources of data.

SECONDARY OUTCOMES:
Genotype-Phenotype Correlation among clinical features and eventual molecular background | 25 years
  Despite the unclear genetic background of Ollier disease and Maffucci syndrome, the secondary outcome aims to correlate genotype and phenotype. This includes, but is not limited to clinical features and genetic background. This will be pursued using the information collected during visits and follow-ups.

OTHER OUTCOMES:
Longitudinal study of disease evolution (including prospective and retrospective data) | 25 years
  This outcome aims to investigate the evolution of Ollier Disease and Maffucci Syndrome during time.
  Main clinical features such as height (cm), number and localization of enchondromas, number and localization of deformities, number and localization of limitations, site/age at malignant transformation will be collected both retrospectively and prospectively in the entire population.
  Those data will be collected both retrospectively and prospectively for all patients via physical examination, clinical reports and imaging.
  An evaluation of these parameters will be performed at each visit to keep track on the progression of the clinical manifestations. Data will be collected to define annualized rate of new clinical manifestations related to age, using analyses such as Kaplan-Meyer and surviving rate.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Sangiorgi, MD, PhD, MS, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Irccs Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Background] Bertucci V, Krafchik BR. What syndrome is this? Ollier disease + vascular lesions: Maffucci syndrome. Pediatr Dermatol. 1995 Mar;12(1):55-8. doi: 10.1111/j.1525-1470.1995.tb00127.x. No abstract available. PMID 7792223
- [Background] Superti-Furga A, Spranger J, Nishimura G. Enchondromatosis revisited: new classification with molecular basis. Am J Med Genet C Semin Med Genet. 2012 Aug 15;160C(3):154-64. doi: 10.1002/ajmg.c.31331. Epub 2012 Jul 12. PMID 22791316
- [Background] Saiji E, Pause FG, Lascombes P, Cerato Biderbost C, Marq NL, Berczy M, Merlini L, Rougemont AL. IDH1 immunohistochemistry reactivity and mosaic IDH1 or IDH2 somatic mutations in pediatric sporadic enchondroma and enchondromatosis. Virchows Arch. 2019 Nov;475(5):625-636. doi: 10.1007/s00428-019-02606-9. Epub 2019 Jun 25. PMID 31240473
- [Background] Pansuriya TC, Kroon HM, Bovee JV. Enchondromatosis: insights on the different subtypes. Int J Clin Exp Pathol. 2010 Jun 26;3(6):557-69. PMID 20661403
- [Background] Herget GW, Strohm P, Rottenburger C, Kontny U, Krauss T, Bohm J, Sudkamp N, Uhl M. Insights into Enchondroma, Enchondromatosis and the risk of secondary Chondrosarcoma. Review of the literature with an emphasis on the clinical behaviour, radiology, malignant transformation and the follow up. Neoplasma. 2014;61(4):365-78. doi: 10.4149/neo_2014_046. PMID 24645839
- [Background] Pansuriya TC, Oosting J, Krenacs T, Taminiau AH, Verdegaal SH, Sangiorgi L, Sciot R, Hogendoorn PC, Szuhai K, Bovee JV. Genome-wide analysis of Ollier disease: Is it all in the genes? Orphanet J Rare Dis. 2011 Jan 14;6:2. doi: 10.1186/1750-1172-6-2. PMID 21235737
- [Background] Silve C, Juppner H. Ollier disease. Orphanet J Rare Dis. 2006 Sep 22;1:37. doi: 10.1186/1750-1172-1-37. PMID 16995932
- [Background] Tsao YP, Tsai CY, Chen WS. Maffucci Syndrome. J Rheumatol. 2015 Dec;42(12):2434-5. doi: 10.3899/jrheum.150216. No abstract available. PMID 26628708
- See also: Institutional webpage of Registries For Rare Hereditary Diseases — https://www.ior.it/en/curarsi-al-rizzoli/registries-rare-hereditary-diseases